CLINICAL TRIAL: NCT03558087
Title: Neoadjuvant Gemcitabine, Cisplatin, Plus Nivolumab in Patients With Muscle-invasive Bladder Cancer With Selective Bladder Sparing
Brief Title: Gemcitabine, Cisplatin, Plus Nivolumab in Patients With Muscle-invasive Bladder Cancer With Selective Bladder Sparing
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Matthew Galsky (Other)
Collaborators: Bristol-Myers Squibb (Industry); Icahn School of Medicine at Mount Sinai (Other)
Responsible Party: Sponsor-Investigator, Matthew Galsky, Sponsor-Investigator, Hoosier Cancer Research Network
Organization: Hoosier Cancer Research Network (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HCRN GU16-257
Record Dates: First submitted 2018-06-05; First posted 2018-06-15 (Actual); Results first posted 2024-06-27 (Actual); Last update posted 2024-06-27 (Actual); Status verified 2024-05

CONDITIONS: Bladder Cancer
Keywords: muscle-invasive
MeSH Terms: conditions — Urinary Bladder Neoplasms | interventions — Nivolumab; Gemcitabine; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Gemcitabine, Cisplatin and Nivolumab (Experimental): Combination Therapy: Nivolumab 360mg IV, Gemcitabine 100mg/m^2 IV ,Cisplatin 70mg/m^2 IV for four 21-day cycles. At restaging, subjects with cT0 or cTa status may undergo cystectomy or continue maintenance Nivolumab 240mg IV for up to 8 14-day cycles. Subjects with > cTa status will undergo cystectomy.
  Interventions: Drug: Nivolumab; Drug: Gemcitabine; Drug: Cisplatin

INTERVENTIONS:
Drug: Nivolumab — Nivolumab 360mg will be administered on Day 1 of each 21 day cycle for four 21-day cycles. Based on response and a balanced patient-physician discussion, subjects may receive nivolumab 240 mg for 8 cycles (cycle = 14 days).
  Other Names: Opdivo
Drug: Gemcitabine — Gemcitabine 1000mg/m^2 will be administered on Days 1 and 8 for four 21-day cycles.
  Other Names: Gemzar
Drug: Cisplatin — Cisplatin 70mg^m2 will be administered on Day 1 for four 21-day cycles.
  Other Names: Platinol

SUMMARY:
This is a phase 2 trial seeking to define the safety and activity of gemcitabine, cisplatin, plus nivolumab as neoadjuvant therapy in patients with muscle-invasive bladder cancer and to define the role of clinical complete response in predicting benefit in patients opting to avoid cystectomy.

ELIGIBILITY:
Inclusion Criteria:

* ECOG Performance Status of ≤ 1 within 28 days prior to registration.
* Histological evidence of clinically localized muscle-invasive urothelial cancer of the bladder (i.e., ct2-4n0m0). candidate for cystectomy as per treating physician.
* Demonstrate adequate organ function per listed criteria:
* Absolute Neutrophil Count (ANC): ≥ 1.5 x 10^9/L
* Hemoglobin (Hgb): ≥ 9 g/dL
* Platelets: ≥ 100 x 10^9/L
* Calculated creatinine clearance: Creatinine ≤ 1.5 or creatinine clearance ≥ 60 mL/min
* Bilirubin: ≤ 1.5 × upper limit of normal (ULN) (except subjects with Gilbert Syndrome, who can have total bilirubin < 3.0 mg/dL)
* Aspartate aminotransferase (AST) : ≤ 3 × ULN
* Alanine aminotransferase (ALT) : ≤ 3 × ULN
* All subjects must have adequate archival tissue identified at screening (i.e., at least 15 unstained slides or paraffin block). Subjects without available archival tissue must be discussed with the sponsor-investigator.
* Women of childbearing potential must have a negative serum or urine pregnancy within 7 days prior to C1D1. NOTE: "Women of childbearing potential" is defined as any female who has experienced menarche and who has not undergone surgical sterilization (hysterectomy or bilateral oophorectomy) or who is not postmenopausal. Menopause is defined clinically as 12 months of amenorrhea in a woman over 45 in the absence of other biological or physiological causes. In addition, women under the age of 62 must have a documented serum follicle stimulating hormone (FSH) level less than 40 mIU/mL.

NOTE: Women of childbearing potential (WOCBP) receiving nivolumab must be willing to abstain from heterosexual intercourse or to use 2 forms of effective methods of contraception from the time of informed consent to 5 months after the last dose of nivolumab or for the timeframe outlined per package insert for chemotherapy. This timeframe also applies to breastfeeding. The two contraception methods can be comprised of two barrier methods, or a barrier method plus a hormonal method. Male subjects capable of fathering a child that are sexually active with partners of childbearing potential must be willing to abstain from heterosexual intercourse or to use 2 forms of effective methods of contraception from the time of informed consent to the timeframe outlined per package insert for chemotherapy. Contraception is not required for nivolumab. The timeframes described in the previous 2 sentences apply to sperm donation. Two contraception methods can be comprised of two barrier methods, or a barrier method plus a hormonal method.

Exclusion Criteria:

* Prior treatment with systemic chemotherapy for muscle-invasive urothelial cancer of the bladder
* Active infection requiring systemic therapy
* Pregnant or breastfeeding (NOTE: breast milk cannot be stored for future use while the mother is being treated on study).
* Any serious or uncontrolled medical disorder that, in the opinion of the investigator, may increase the risk associated with study participation or study drug administration, impair the ability of the subject to receive protocol therapy, or interfere with the interpretation of study results.
* Prior malignancy active within the previous 3 years except for locally curable cancers that have been apparently cured.
* Subjects with active, known or suspected autoimmune disease. Subjects with vitiligo, type I diabetes mellitus, residual hypothyroidism due to autoimmune condition only requiring hormone replacement, psoriasis not requiring systemic treatment, or conditions not expected to recur in the absence of an external trigger are permitted to enroll.
* Subjects with a condition requiring systemic treatment with either corticosteroids (> 10 mg daily prednisone equivalents) or other immunosuppressive medications within 14 days of study drug administration. Inhaled or topical steroids and adrenal replacement doses > 10 mg daily prednisone equivalents are permitted in the absence of active autoimmune disease.
* Prior treatment with an anti-PD-1, anti-PD-L1, anti-PD-L2, anti-CTLA-4 antibody, or any other antibody or drug specifically targeting T-cell co-stimulation or immune checkpoint pathways.
* Grade ≥ 2 neuropathy (NCI CTCAE version 4).
* Prior radiation therapy for bladder cancer
* Positive test for hepatitis B virus surface antigen (HBV sAg) or hepatitis C virus ribonucleic acid (RNA) or hepatitis C antibody (HCV antibody) indicating acute or chronic infection.
* Known history of testing positive for human immunodeficiency virus (HIV) or known acquired immunodeficiency syndrome (AIDS).
* Evidence of interstitial lung disease or active, non-infectious pneumonitis.
* Solid organ or allogeneic stem cell transplant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2018-07-13 (Actual); Primary Completion 2024-02-16 (Actual); Study Completion 2024-03-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Galsky, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (7):
- United States (7):
  - City of Hope, Duarte, California
  - Univerity of Southern California, Los Angeles, California
  - Icahn School of Medicine: Tisch Cancer Institute at Mount Sinai Medical Center, New York, New York
  - Oregon Health & Science University, Portland, Oregon
  - Penn Medicine Abramson Cancer Center, Philadelphia, Pennsylvania
  - Huntsman Cancer Institute University of Utah, Salt Lake City, Utah
  - University of Wisconsin, Madison, Wisconsin

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Gemcitabine, Cisplatin and Nivolumab
Started | 76
Completed | 76
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Gemcitabine, Cisplatin and Nivolumab
Number analyzed (Participants) | 76
Age, Continuous [Median (Full Range); unit: years] | 69 [39 to 85]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16
  Male | 60
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 9
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 58
  More than one race | 0
  Unknown or Not Reported | 8
Region of Enrollment [Number; unit: participants]
  United States | 76
Clinical stage [Count of Participants; unit: Participants] — Tumor Node Metastasis (TNM) Staging. This system classifies tumors by size and extent of the primary tumor (T), involvement of regional lymph nodes (N), and the presence or absence of distant metastases (M).
  T0=No evidence of primary tumor, Tis=Carcinoma in situ, and T1, T2, T3, T4=Increasing size and/or local extension of the primary tumor, TX=Not assessed.
  N0=No Regional lymph node metastases, N1, N2, N3=Increasing number or extent of regional lymph node involvement, NX=not assessed.
  M0=No distant metastases, M1=Distant metastases present
  Participants
    cT2N0M0 | 43
    cT3N0M0 | 24
    cT4N0M0 | 9
Histology [Count of Participants; unit: Participants]
  Urothelial Cancer (UC) | 57
  UC with squamous | 7
  UC with glandular | 2
  UC with micropapillary | 6
  UC with other variant | 4

OUTCOME MEASURES:

1. Primary Outcome: Clinical Complete Response (CCR) Rate
Description: Clinical complete response rate will be defined as the percentage of patients who achieved cT0 or cTa disease after gemcitabine, cisplatin, plus nivolumab.
Time Frame: 24 months
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Gemcitabine, Cisplatin and Nivolumab
Number analyzed (Participants) | 76
Percentage of participants | 43 [32 to 55]

2. Primary Outcome: Predict Benefit From Treatment
Description: Determine the ability of clinical complete response (cT0 or cTa) to predict benefit from treatment.Benefit will be defined as a pathologic complete response (<pT1) in patients undergoing cystectomy and 2 year metastasis-free in patients pursuing surveillance.
  The positive predictive value of CCR with 95% confidence interval are presented in Outcome Measure Data Table. Positive predictive value is the ratio of patients truly diagnosed as positive to all those who had positive test results.
Time Frame: 24 months
Population: Among the 33 patients achieving a CCR, only one opted for immediate cystectomy with surgical pathology, revealing a low-grade ypTaN0 urothelial cancer (UC). Therefore 32 patients were used for this outcome measure.
Measure: Number (95% Confidence Interval); unit: Proportion of CCR patients
Arm/Group | Gemcitabine, Cisplatin and Nivolumab
Number analyzed (Participants) | 32
Proportion of CCR patients | 0.97 [0.91 to 1]

3. Secondary Outcome: Adverse Events
Description: The frequency and severity of all grade 3+ treatment-emergent adverse events occurring in at least 10% of patients are reported by CTCAEv4 term and grade.
Time Frame: AE had been recorded from time of signed informed consent until 100 days after discontinuation of study drug(s) or until a new anti-cancer treatment starts, whichever occurs first, up to a maximum of 13 months.
Measure: Number; unit: participants
Arm/Group | Gemcitabine, Cisplatin and Nivolumab
Number analyzed (Participants) | 76
participants
  ANEMIA | 12
  NEUTROPHIL COUNT DECREASED | 26
  URINARY TRACT INFECTION | 13
  HYPONATREMIA | 5
  HYPERTENSION | 4
  WHITE BLOOD CELL DECREASED | 3
  PLATELET COUNT DECREASED | 4
  HEMATURIA | 3
  DYSPNEA | 1
  VOMITING | 1
  ABDOMINAL PAIN | 2
  HYPOKALEMIA | 3
  PAIN | 1
  ASPARTATE AMINOTRANSFERASE INCREASED | 1
  DEPRESSION | 1
  ANXIETY | 1
  HYPERGLYCEMIA | 2

4. Secondary Outcome: Bladder Intact Overall Survival
Description: Bladder-intact overall survival is defined as the time from initiation of treatment until death or cystectomy.
Time Frame: Up to a maximum of 60 months
Population: Bladder-intact overall survival results are showing in accordance with CCR status. Out of 76 patients, 33 patients achieved a clinical complete response, and 43 patients did not achieve a clinical complete response.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Gemcitabine, Cisplatin and Nivolumab
Number analyzed (Participants) | 76
Months
  CCR Patients: number analyzed (Participants) | 33
  CCR Patients | NA [47.34 to NA] — Not enough events occur to calculate the median and upper 95% confidence interval
  Non-CCR Patients: number analyzed (Participants) | 43
  Non-CCR Patients | 4.53 [4.24 to 4.93]

5. Secondary Outcome: Recurrence-free Survival
Description: Recurrence-free survival is defined as the time from initiation of treatment to death or recurrence, depending on which occurs first
Time Frame: Up to a maximum of 60 months
Population: Recurrence-free survival results are showing in accordance with CCR status. Out of 76 patients, 33 patients achieved a clinical complete response, and 43 patients did not achieve a clinical complete response.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Gemcitabine, Cisplatin and Nivolumab
Number analyzed (Participants) | 76
Months
  CCR Patients: number analyzed (Participants) | 33
  CCR Patients | 51.52 [39.92 to NA] — Not enough events occur to calculate the upper 95% confidence interval.
  Non-CCR Patients: number analyzed (Participants) | 43
  Non-CCR Patients | NA [24.21 to NA] — Not enough events occur to calculate the median and upper 95% confidence interval.

6. Secondary Outcome: Pathologic Complete Response Rate in Patients Undergoing Cystectomy
Description: Pathologic complete response rate in patients undergoing radical cystectomy is defined as the proportion of patients with <pT1
Time Frame: Up to a maximum of 53 months
Population: Only 8 patients achieving a clinical complete response (CCR) later underwent cystectomy, and 34 patients not achieving a CCR underwent cystectomy.
Measure: Count of Participants; unit: Participants
Arm/Group | Gemcitabine, Cisplatin and Nivolumab
Number analyzed (Participants) | 42
Participants
  CCR Patients: number analyzed (Participants) | 8
  CCR Patients | 1
  Non-CCR Patients: number analyzed (Participants) | 34
  Non-CCR Patients | 3

7. Secondary Outcome: Association Between a Prespecified Panel of Genomic Biomarkers and Benefit From Treatment in Patients Achieving a Clinical Complete Response.
Description: Benefit will be defined as a pathologic complete response (p<T1) in patients undergoing cystectomy and 2 years metastasis-free in patients pursuing surveillance.
  The positive predictive value of CCR with or without genomic alterations in baseline TURBT tissue for a composite outcome measure of 2-year bladder-intact survival in patients forgoing immediate cystectomy or <ypT1N0 in patients undergoing immediate cystectomy are presented with 95% confidence interval in Outcome Measure Data Table.
  Positive predictive value is the ratio of patients truly diagnosed as positive to all those who had positive test results.
Time Frame: 24 months
Measure: Number (95% Confidence Interval); unit: Proportion of CCR patients
Arm/Group | Gemcitabine, Cisplatin and Nivolumab
Number analyzed (Participants) | 33
Proportion of CCR patients | 0.72 [0.56 to 0.87]

8. Secondary Outcome: Overall Survival
Description: Overall survival is defined as the time from initiation of treatment to death.
Time Frame: Up to a maximum of 60 months
Population: Overall survival results are showing in accordance with CCR status. Out of 76 patients, 33 patients achieved a clinical complete response, and 43 patients did not achieve a clinical complete response.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Gemcitabine, Cisplatin and Nivolumab
Number analyzed (Participants) | 76
Months
  CCR Patients: number analyzed (Participants) | 33
  CCR Patients | NA [NA to NA] — Not enough events occur to calculate the median and 95% confidence interval.
  Non-CCR Patients: number analyzed (Participants) | 43
  Non-CCR Patients | NA [41.49 to NA] — Not enough events occur to calculate the median and upper 95% confidence interval.

ADVERSE EVENTS:
Time Frame: All-Cause Mortality was monitored up to a maximum of 60 months. Serious Adverse Events and Other (Not Including Serious) Adverse Events were monitored up to 13 months.
Arm/Group | Gemcitabine, Cisplatin and Nivolumab
All-Cause Mortality (participants affected / at risk) | 13/76
Serious Adverse Events (participants affected / at risk) | 40/76
Other Adverse Events (participants affected / at risk) | 76/76
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Gemcitabine, Cisplatin and Nivolumab (N=76)
ABDOMINAL PAIN (Gastrointestinal disorders) | 2 (2)
ACUTE KIDNEY INJURY (Renal and urinary disorders) | 5 (5)
ADRENAL INSUFFICIENCY (Endocrine disorders) | 1 (1)
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 1 (1)
ANEMIA (Blood and lymphatic system disorders) | 1 (2)
ATRIAL FIBRILLATION (Cardiac disorders) | 2 (2)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 1 (1)
BLOOD AND LYMPHATIC SYSTEM DISORDERS - OTHER, SPECIFY (Blood and lymphatic system disorders) | 1 (1)
BLOOD BILIRUBIN INCREASED (Investigations) | 1 (1)
DEPRESSION (Psychiatric disorders) | 1 (1)
DYSPNEA (Respiratory, thoracic and mediastinal disorders) | 1 (2)
FEBRILE NEUTROPENIA (Blood and lymphatic system disorders) | 1 (1)
FEVER (General disorders) | 1 (1)
HEMATURIA (Renal and urinary disorders) | 1 (1)
HYPERTHYROIDISM (Endocrine disorders) | 1 (1)
HYPONATREMIA (Metabolism and nutrition disorders) | 4 (4)
HYPOTENSION (Vascular disorders) | 1 (1)
INFECTIONS AND INFESTATIONS - OTHER, SPECIFY (Infections and infestations) | 3 (4)
KIDNEY INFECTION (Infections and infestations) | 1 (1)
LUNG INFECTION (Infections and infestations) | 1 (1)
PLATELET COUNT DECREASED (Investigations) | 1 (1)
RENAL AND URINARY DISORDERS - OTHER, SPECIFY (Renal and urinary disorders) | 2 (3)
SEPSIS (Infections and infestations) | 4 (6)
SMALL INTESTINAL OBSTRUCTION (Gastrointestinal disorders) | 1 (1)
STROKE (Nervous system disorders) | 1 (1)
THROMBOEMBOLIC EVENT (Vascular disorders) | 3 (3)
URINARY TRACT INFECTION (Infections and infestations) | 10 (11)
VOMITING (Gastrointestinal disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Gemcitabine, Cisplatin and Nivolumab (N=76)
ABDOMINAL DISTENSION (Gastrointestinal disorders) | 1 (1)
ABDOMINAL PAIN (Gastrointestinal disorders) | 8 (10)
ACTIVATED PARTIAL THROMBOPLASTIN TIME PROLONGED (Investigations) | 2 (2)
ACUTE KIDNEY INJURY (Renal and urinary disorders) | 3 (5)
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 10 (17)
ALKALINE PHOSPHATASE INCREASED (Investigations) | 5 (6)
ALOPECIA (Skin and subcutaneous tissue disorders) | 20 (20)
ANEMIA (Blood and lymphatic system disorders) | 52 (146)
ANKLE FRACTURE (Injury, poisoning and procedural complications) | 1 (1)
ANOREXIA (Metabolism and nutrition disorders) | 22 (25)
ANXIETY (Psychiatric disorders) | 5 (6)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 1 (1)
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 9 (21)
ATELECTASIS (Respiratory, thoracic and mediastinal disorders) | 1 (1)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 13 (14)
BLOATING (Gastrointestinal disorders) | 3 (5)
BLOOD AND LYMPHATIC SYSTEM DISORDERS - OTHER, SPECIFY (Blood and lymphatic system disorders) | 16 (27)
BLOOD BILIRUBIN INCREASED (Investigations) | 2 (3)
BLURRED VISION (Eye disorders) | 4 (6)
BONE PAIN (Musculoskeletal and connective tissue disorders) | 1 (1)
BURN (Injury, poisoning and procedural complications) | 1 (1)
CHILLS (General disorders) | 2 (2)
CHOLESTEROL HIGH (Investigations) | 4 (4)
COGNITIVE DISTURBANCE (Nervous system disorders) | 1 (1)
COLITIS (Gastrointestinal disorders) | 1 (1)
CONSTIPATION (Gastrointestinal disorders) | 35 (38)
COUGH (Respiratory, thoracic and mediastinal disorders) | 6 (6)
CREATININE INCREASED (Investigations) | 36 (64)
CYSTITIS NONINFECTIVE (Renal and urinary disorders) | 1 (1)
DEHYDRATION (Metabolism and nutrition disorders) | 3 (4)
DEPRESSION (Psychiatric disorders) | 5 (7)
DIARRHEA (Gastrointestinal disorders) | 11 (14)
DIZZINESS (Nervous system disorders) | 7 (9)
DRY MOUTH (Gastrointestinal disorders) | 2 (2)
DRY SKIN (Skin and subcutaneous tissue disorders) | 3 (3)
DYSGEUSIA (Nervous system disorders) | 9 (9)
DYSPEPSIA (Gastrointestinal disorders) | 1 (1)
DYSPNEA (Respiratory, thoracic and mediastinal disorders) | 19 (24)
EAR AND LABYRINTH DISORDERS - OTHER, SPECIFY (Ear and labyrinth disorders) | 1 (1)
EAR PAIN (Ear and labyrinth disorders) | 1 (1)
EDEMA LIMBS (General disorders) | 8 (12)
ENDOCRINE DISORDERS - OTHER, SPECIFY (Endocrine disorders) | 2 (2)
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 4 (4)
EYE DISORDERS - OTHER, SPECIFY (Eye disorders) | 1 (1)
FACIAL PAIN (General disorders) | 1 (1)
FALL (Injury, poisoning and procedural complications) | 3 (5)
FATIGUE (General disorders) | 54 (80)
FEVER (General disorders) | 4 (5)
FLANK PAIN (Musculoskeletal and connective tissue disorders) | 1 (1)
FLASHING LIGHTS (Eye disorders) | 1 (1)
FLATULENCE (Gastrointestinal disorders) | 1 (1)
FLU LIKE SYMPTOMS (General disorders) | 1 (1)
FLUSHING (Vascular disorders) | 2 (2)
GAIT DISTURBANCE (General disorders) | 2 (2)
GASTROESOPHAGEAL REFLUX DISEASE (Gastrointestinal disorders) | 3 (3)
GASTROINTESTINAL DISORDERS - OTHER, SPECIFY (Gastrointestinal disorders) | 5 (6)
GENERAL DISORDERS AND ADMINISTRATION SITE CONDITIONS - OTHER, SPECIFY (General disorders) | 6 (8)
GENERALIZED MUSCLE WEAKNESS (Musculoskeletal and connective tissue disorders) | 3 (4)
GGT INCREASED (Investigations) | 1 (1)
HEADACHE (Nervous system disorders) | 10 (12)
HEARING IMPAIRED (Ear and labyrinth disorders) | 2 (2)
HEMATOMA (Vascular disorders) | 1 (1)
HEMATURIA (Renal and urinary disorders) | 19 (26)
HEMORRHOIDS (Gastrointestinal disorders) | 1 (1)
HEPATOBILIARY DISORDERS - OTHER, SPECIFY (Hepatobiliary disorders) | 1 (1)
HICCUPS (Respiratory, thoracic and mediastinal disorders) | 2 (2)
HOARSENESS (Respiratory, thoracic and mediastinal disorders) | 2 (3)
HYPERCALCEMIA (Metabolism and nutrition disorders) | 1 (1)
HYPERGLYCEMIA (Metabolism and nutrition disorders) | 32 (57)
HYPERKALEMIA (Metabolism and nutrition disorders) | 8 (12)
HYPERMAGNESEMIA (Metabolism and nutrition disorders) | 2 (2)
HYPERNATREMIA (Metabolism and nutrition disorders) | 1 (1)
HYPERTENSION (Vascular disorders) | 16 (28)
HYPERTHYROIDISM (Endocrine disorders) | 3 (5)
HYPERTRIGLYCERIDEMIA (Metabolism and nutrition disorders) | 1 (1)
HYPERURICEMIA (Metabolism and nutrition disorders) | 3 (3)
HYPOALBUMINEMIA (Metabolism and nutrition disorders) | 12 (18)
HYPOCALCEMIA (Metabolism and nutrition disorders) | 11 (18)
HYPOGLYCEMIA (Metabolism and nutrition disorders) | 3 (5)
HYPOKALEMIA (Metabolism and nutrition disorders) | 12 (15)
HYPOMAGNESEMIA (Metabolism and nutrition disorders) | 14 (29)
HYPONATREMIA (Metabolism and nutrition disorders) | 20 (47)
HYPOPHOSPHATEMIA (Metabolism and nutrition disorders) | 4 (6)
HYPOTENSION (Vascular disorders) | 3 (5)
HYPOTHYROIDISM (Endocrine disorders) | 2 (2)
HYPOXIA (Respiratory, thoracic and mediastinal disorders) | 1 (3)
ILEUS (Gastrointestinal disorders) | 2 (2)
IMMUNE SYSTEM DISORDERS - OTHER, SPECIFY (Immune system disorders) | 1 (1)
INFECTIONS AND INFESTATIONS - OTHER, SPECIFY (Infections and infestations) | 3 (3)
INFUSION RELATED REACTION (General disorders) | 2 (4)
INFUSION SITE EXTRAVASATION (General disorders) | 1 (1)
INJECTION SITE REACTION (General disorders) | 3 (3)
INSOMNIA (Psychiatric disorders) | 9 (9)
INVESTIGATIONS - OTHER, SPECIFY (Investigations) | 3 (4)
KIDNEY INFECTION (Infections and infestations) | 1 (1)
LEFT VENTRICULAR SYSTOLIC DYSFUNCTION (Cardiac disorders) | 1 (1)
LIBIDO DECREASED (Psychiatric disorders) | 1 (1)
LIPASE INCREASED (Investigations) | 5 (9)
LOCALIZED EDEMA (General disorders) | 1 (1)
LYMPHOCYTE COUNT DECREASED (Investigations) | 4 (4)
MEMORY IMPAIRMENT (Nervous system disorders) | 1 (1)
METABOLISM AND NUTRITION DISORDERS - OTHER, SPECIFY (Metabolism and nutrition disorders) | 7 (17)
MUCOSITIS ORAL (Gastrointestinal disorders) | 2 (2)
MUSCLE WEAKNESS UPPER LIMB (Musculoskeletal and connective tissue disorders) | 1 (2)
MUSCULOSKELETAL AND CONNECTIVE TISSUE DISORDER - OTHER, SPECIFY (Musculoskeletal and connective tissue disorders) | 3 (3)
NASAL CONGESTION (Respiratory, thoracic and mediastinal disorders) | 3 (3)
NAUSEA (Gastrointestinal disorders) | 43 (58)
NECK PAIN (Musculoskeletal and connective tissue disorders) | 1 (2)
NERVOUS SYSTEM DISORDERS - OTHER, SPECIFY (Nervous system disorders) | 1 (1)
NEURALGIA (Nervous system disorders) | 1 (2)
NEUTROPHIL COUNT DECREASED (Investigations) | 52 (151)
NON-CARDIAC CHEST PAIN (General disorders) | 1 (1)
ORAL PAIN (Gastrointestinal disorders) | 1 (1)
PAIN (General disorders) | 8 (13)
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 4 (4)
PALPITATIONS (Cardiac disorders) | 1 (1)
PAPULOPUSTULAR RASH (Infections and infestations) | 1 (1)
PARESTHESIA (Nervous system disorders) | 1 (1)
PELVIC PAIN (Reproductive system and breast disorders) | 1 (1)
PERINEAL PAIN (Reproductive system and breast disorders) | 1 (4)
PERIORBITAL EDEMA (Skin and subcutaneous tissue disorders) | 1 (1)
PERIORBITAL INFECTION (Infections and infestations) | 1 (1)
PERIPHERAL MOTOR NEUROPATHY (Nervous system disorders) | 1 (3)
PERIPHERAL SENSORY NEUROPATHY (Nervous system disorders) | 6 (6)
PHLEBITIS (Vascular disorders) | 2 (2)
PHOTOSENSITIVITY (Skin and subcutaneous tissue disorders) | 1 (1)
PLATELET COUNT DECREASED (Investigations) | 29 (59)
PRESYNCOPE (Nervous system disorders) | 2 (2)
PRODUCTIVE COUGH (Respiratory, thoracic and mediastinal disorders) | 2 (2)
PROTEINURIA (Renal and urinary disorders) | 9 (10)
PRURITUS (Skin and subcutaneous tissue disorders) | 11 (13)
PSYCHIATRIC DISORDERS - OTHER, SPECIFY (Psychiatric disorders) | 1 (1)
RASH ACNEIFORM (Skin and subcutaneous tissue disorders) | 3 (3)
RASH MACULO-PAPULAR (Skin and subcutaneous tissue disorders) | 13 (14)
RENAL AND URINARY DISORDERS - OTHER, SPECIFY (Renal and urinary disorders) | 18 (26)
RESPIRATORY, THORACIC AND MEDIASTINAL DISORDERS - OTHER, SPECIFY (Respiratory, thoracic and mediastinal disorders) | 3 (3)
SEPSIS (Infections and infestations) | 1 (1)
SEROMA (Injury, poisoning and procedural complications) | 1 (1)
SERUM AMYLASE INCREASED (Investigations) | 7 (15)
SINUS DISORDER (Respiratory, thoracic and mediastinal disorders) | 1 (1)
SINUS TACHYCARDIA (Cardiac disorders) | 2 (2)
SINUSITIS (Infections and infestations) | 1 (1)
SKIN AND SUBCUTANEOUS TISSUE DISORDERS - OTHER, SPECIFY (Skin and subcutaneous tissue disorders) | 10 (13)
SOMNOLENCE (Nervous system disorders) | 1 (1)
SORE THROAT (Respiratory, thoracic and mediastinal disorders) | 1 (1)
STOMA SITE INFECTION (Infections and infestations) | 2 (2)
SUPERFICIAL THROMBOPHLEBITIS (Vascular disorders) | 3 (3)
SURGICAL AND MEDICAL PROCEDURES - OTHER, SPECIFY (Surgical and medical procedures) | 2 (2)
SYNCOPE (Nervous system disorders) | 2 (3)
THROMBOEMBOLIC EVENT (Vascular disorders) | 2 (2)
TINNITUS (Ear and labyrinth disorders) | 21 (22)
TOOTHACHE (Gastrointestinal disorders) | 3 (3)
TREMOR (Nervous system disorders) | 4 (5)
UPPER RESPIRATORY INFECTION (Infections and infestations) | 2 (2)
URINARY FREQUENCY (Renal and urinary disorders) | 7 (7)
URINARY INCONTINENCE (Renal and urinary disorders) | 2 (2)
URINARY RETENTION (Renal and urinary disorders) | 1 (1)
URINARY TRACT INFECTION (Infections and infestations) | 15 (29)
URINARY TRACT PAIN (Renal and urinary disorders) | 8 (12)
URINARY URGENCY (Renal and urinary disorders) | 4 (4)
UROSTOMY LEAK (Injury, poisoning and procedural complications) | 1 (1)
VASCULAR DISORDERS - OTHER, SPECIFY (Vascular disorders) | 1 (1)
VERTIGO (Ear and labyrinth disorders) | 1 (1)
VESTIBULAR DISORDER (Ear and labyrinth disorders) | 1 (1)
VOMITING (Gastrointestinal disorders) | 14 (19)
WATERING EYES (Eye disorders) | 1 (2)
WEIGHT GAIN (Investigations) | 2 (4)
WEIGHT LOSS (Investigations) | 10 (15)
WHITE BLOOD CELL DECREASED (Investigations) | 31 (65)
WOUND INFECTION (Infections and infestations) | 1 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-08-12): https://cdn.clinicaltrials.gov/large-docs/87/NCT03558087/Prot_SAP_000.pdf